CLINICAL TRIAL: NCT01627262
Title: Double-blind, Randomised, Placebo-controlled, Parallel-group, Multi-centre Phase III Clinical Study on the Efficacy and Tolerability of Mesalazine Pellets vs. Placebo in Diverticular Disease
Brief Title: Mesalamine for Uncomplicated Diverticular Disease: a Randomized, Double-blind, Placebo-controlled Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAG-20/DIV
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Colonic Diverticulosis
Keywords: diverticular disease; colonic diverticulosis; mesalamine; placebo; randomized
MeSH Terms: conditions — Diverticulosis, Colonic; Diverticular Diseases | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Mesalamine (Experimental)
  Interventions: Drug: Mesalamine

INTERVENTIONS:
Drug: Mesalamine — 3x1000mg mesalamine granules per day
  Other Names: Salofalk granules
  Arms: Mesalamine
Drug: Placebo — 3x1000mg placebo granules per day
  Other Names: Placebo granules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether mesalamine is effective in the treatment of uncomplicated diverticular disease by reducing the pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diverticular disease with acute pain without serious complications
* Lower abdominal pain of moderate or severe intensity at least during the last 4 days before study inclusion

Exclusion Criteria:

* Chronic inflammatory bowel disease
* Fever or other signs of serious complications.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2002-05; Primary Completion 2004-08 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The change in intensity of lower abdominal pain during the first four weeks of treatment (SPID 0-28) | 4 weeks
  The change in intensity of lower abdominal pain during the first four weeks of treatment, defined as the cumulative difference of the daily pain intensity score from the first day of study medication intake (day 1) to week 4

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kruis, MD, Principal Investigator — Ev. Krankenhaus Kalk, University of Cologne
Locations (1):
- Ev. Krankenhaus Kalk, University of Cologne, Cologne, Germany

REFERENCES:
- [Result] Kruis W, Meier E, Schumacher M, Mickisch O, Greinwald R, Mueller R; German SAG-20 Study Group. Randomised clinical trial: mesalazine (Salofalk granules) for uncomplicated diverticular disease of the colon--a placebo-controlled study. Aliment Pharmacol Ther. 2013 Apr;37(7):680-90. doi: 10.1111/apt.12248. Epub 2013 Feb 17. PMID 23414061